CLINICAL TRIAL: NCT05636878
Title: Creation and Evaluation of a Mobile Intervention Team in Perinatal Psychiatry (0-3 Years) in Meurthe-et-Moselle Sud
Acronym: EMPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RIPH 2021-06; 2021-A02678-33 (Other: ANSM)
Record Dates: First submitted 2022-09-14; First posted 2022-12-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-12

CONDITIONS: Abnormality
Keywords: Perinatal; Psychiatry; psychomoteur; children
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: For the primary objective, i.e., analysis of the effect of the intervention at age 2 (and the first SO, i.e., analysis of the effect of the intervention at age 4), a difference-in-differences analysis will be performed. That is, the difference in the prevalence of abnormal psychomotor development at age 2 (and at age 4) before and after the implementation of the EMPPer in the target territory will be compared to the difference in the prevalence of abnormal psychomotor development at age 2 (and at age 4) between the periods corresponding to the implementation of the EMPPer in the territories that did not benefit from it, using a mixed linear regression model with psychomotor developmental abnormalities as the variable to be explained, year (pre vs. post intervention) and region (with vs. without intervention) as explanatory variables, and which will include the year*region interaction. The assumption of equivalence of temporal developmental trends here and elsewhere will be tested
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With EMPPer (Experimental): All children (0 to 3 years old) in the areas Meurthe-et-Moselle South will benefit from the intervention of the Mobile Perinatal Psychiatry Team (EMPPer)
  Interventions: Other: Mobile Intervention Team in Perinatal Psychiatry (EMPPer)
- without EMPPer (No Intervention): All children (0 to 3 years) from Strasbourg and Reims will not benefit from the Mobile Intervention Team in Perinatal Psychiatry

INTERVENTIONS:
Other: Mobile Intervention Team in Perinatal Psychiatry (EMPPer) — The Mobile Intervention Team in Perinatal Psychiatry consists in going towards the most excluded patients, changing the organization of care compared to the current practice and facilitating access to care for the most vulnerable populations
  Arms: With EMPPer

SUMMARY:
The research system is a Mobile Perinatal Psychiatry Team (EMPPer), for children aged 0 to 3 and their parents. it facilitates access to psychiatric care by going to families who need it and who are in difficulty to ensure this process.

This device, already deployed in a dozen French cities for several years, convinced the teams of its interest, without demonstrating its effectiveness by evaluation conducted according to research standards. The deployment of a Mobile Perinatal Psychiatry Team in a region not yet equipped (Meurthe-et-Moselle Sud) would therefore offer the opportunity to assess its effectiveness,

The main objective of the research is to evaluate the effect of the EMPPer on the prevalence of abnormalities in the psychomotor development of children at the age of 2 years, in comparison with similar territories that do not benefit from it, and in comparison with the period preceding the establishment of the EMPPer in the targeted territory.

DETAILED DESCRIPTION:
Context:

The inflation of psycho-social vulnerability and precariousness situations, of parents or isolated mothers with their young child, who do not have easy access to perinatal psychiatry care structures, incites us to develop a modality of home interventions. This is part of a therapeutic perspective of the parenting process and parent-child interactions and a preventive perspective of the child's development. This system is a Mobile Perinatal Psychiatry Team and is also designed for professionals working in early childhood (such as the homes that take in parents). They are in demand for direct interventions with patients, but also indirect interventions, for assistance in the detection of early disorders in children and for referral to psychiatric care.

The main objective of the research is to evaluate the effect of the EMPPer on the prevalence of abnormalities in the psychomotor development of children at the age of 2 years , in comparison with similar territories that do not benefit from it, and in comparison with the period before the EMPPer was implemented in the targeted territory.

The secondary objectives are:

* to evaluate the long-term effect of the EMPPer on the prevalence of child language delay at age 4, compared with similar territories without the EMPPer and compared with the period before the EMPPer was implemented in the target territory
* to evaluate the EMPPer implementation process, in terms of context, interventions implemented, implementation, and impact mechanisms
* to evaluate the medico-economic impact at 2 years of the implementation of the EMPPer.

Methodology:

EMPER is a quasi-experimental study combining a before-and-after EMPPer implementation design with a here-and-now design. A concomitant process evaluation will also be conducted to assess the actual implementation of the intervention, the impact mechanisms of the intervention on the judgment criteria, and to understand precisely the context of implementation in order to better identify the transferability and sustainability of the intervention.

the study will include all the children of the EMPPer sector as well as those of the Reims and Strasbourg hospital sectors. Data from their 24th month and 3-4 years examinations will be collected .

Process evaluation will be based on mixed methods.It will be based on standardized data collection using an observation book and validated measurement instruments such as the satisfaction and therapeutic alliance questionnaire. It will include all users and professionals involved in the implementation of the EMPPer and willing to participate.

The qualitative approach will make it possible, through field observations and semi-structured interviews with professionals and volunteer users, to specify certain elements relating to the intervention itself, such as the organizations within the EMPPer, but also its implementation (possible adaptations of the intervention) or its impact mechanisms.

Expected results are that the deployment of an EMPPer will allow:

* To promote early detection of interaction disorders in order to limit theirs consequences on somatic, cognitive and psychomotor development
* To promote early detection of neurodevelopmental disorders
* To promote early intervention, in connection with early childhood partners
* To facilitate the care pathway of the young patient and his family by allowing easier access to care.

ELIGIBILITY:
Inclusion Criteria:

* Children benefiting from EMPPer intervention
* Children affiliated or entitled to a social security system
* Children for whom the holder of parental authority has received informed information about the study and has co-signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

* Children whose parents are visiting the region ( vacations, family visits ...)
* Children for whom the 2 holders of parental authority do not speak french
* Children for whom both parents do not know how to read

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4260 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-08-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with anomaly of the child's psychomotor development at age 2 years | up to 24 months
  It defined by the fact of having at least one box ticked "no" in the psychomotor development section of the medical part of the third health certificate , carried out after a systematic examination at the age of 24 months of the child

SECONDARY OUTCOMES:
Number of Children with Language Delay at age 4 | up to 4 years
  It evaluated during a health examination systematically carried out at the age of 4 years for the child attending school
Therapeutic alliance score | up to 4 years
  Therapeutic alliance score (parents of the child) on the Working Alliance Inventory questionnaire (Bottemine, 2017; Horvath 1989)
User satisfaction score | up to 4 years
  using the questionnaire offered to parents of children in care by the Nancy Psychotherapy Center as part of its quality approach
the cost of care for children with a psychomotor development problem | 2 years
  it makes it possible to carry out a medico-economic analysis, and to estimate the difference in costs between the two strategies of care (with and without EMPPer)

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne LIGIER, Pr., Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapique de Nancy, Laxou, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antenatal and postnatal mental health: clinical management and service guidance. London: National Institute for Health and Care Excellence (NICE); 2018 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK553127/ PMID 31990493
- [Background] Alla F, Guillemin F, Colombo MC, Roy B, Maeder C. [Diagnostic value of ERTL4: a screening test of language disorders in 4-year-old children]. Arch Pediatr. 1998 Oct;5(10):1082-8. doi: 10.1016/s0929-693x(99)80004-9. French. PMID 9809150
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Dupont C, Touzet S, Ploin D, Croidieu C, Balsan M, Mazas AS, Rudigoz RC. [Evaluation of the perinatal network professionals' integration: study about 653 professionals of AURORE network]. J Gynecol Obstet Biol Reprod (Paris). 2007 Jun;36(4):375-83. doi: 10.1016/j.jgyn.2007.01.003. Epub 2007 Feb 20. French. PMID 17317036